CLINICAL TRIAL: NCT06693037
Title: A Cohort Study of Different Choice of Adjuvant Therapy in Non-PCR Patients With HER2 Positive Early Breast Cancer After Neoadjuvant Therapy
Brief Title: Adjuvant Therapy Choice for Non-pCR HER2 Positive Early Breast Cancer After Neoadjuvant Therapy
Acronym: nonPHER
Status: Recruiting | Type: Observational
Sponsor: Shu Wang (Other)
Responsible Party: Sponsor-Investigator, Shu Wang, director of breast center, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Other Study IDs: PKUPH2024Z169
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: HER2-positive Breast Cancer
Keywords: neoadjuvant chemotherapy; non-pCR; T-DM1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Tumor paraffin sample for each patient
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trastuzumab combined with pertuzumab: The postoperative adjuvant regimen was trastuzumab combined with pertuzumab, and the planned treatment duration was 1 year
- T-DM1: The postoperative adjuvant regimen was T-DM1, and the planned treatment duration was 1 year

SUMMARY:
Chemotherapy combined with trastuzumab and patuzumab is the standard neoadjuvant therapy for HER2 positive breast cancer patients. The survival rate of patients with pathological complete response (PCR) after neoadjuvant therapy was significantly better than that of patients with tumor residue, that is, non-PCR. Therefore, studies have confirmed that adjuvant therapy for patients with non-PCR after neoadjuvant chemotherapy can further improve the prognosis and survival of this population. However, the results of previous studies are based on trastuzumab target therapy in neoadjuvant therapy. Therefore, there are different recommendations for the current guidelines of adjuvant therapy after trastuzumab combined pertuzumab target neoadjuvant therapy. Patients with HER2 positive breast cancer who received trastuzumab and patuzumab based neoadjuvant therapy had invasive residual cancer in postoperative pathology. The effect of postoperative adjuvant therapy with trastuzumab and patuzumab or replacement of T-DM1 on survival.

DETAILED DESCRIPTION:
Investigators retrospectively recruited patients with HER2 positive breast cancer who received trastuzumab and patuzumab based neoadjuvant therapy had invasive residual cancer in postoperative pathology from January 1, 2019 to November 31, 2024, and prospectively recruit patients of the same type from December 1, 2024 to December 31, 2028.

Inclusion Criteria:

1. Patients with HER2 positive breast cancer were diagnosed by biopsy in Peking University People's hospital;
2. The clinical stages before treatment were T1-T4, N0-N3, M0;
3. Received treatment and operation in our hospital, and had hospitalization records;
4. Receive at least 4 cycles of trastuzumab and pertuzumab target therapy combined chemotherapy as neoadjuvant therapy
5. Postoperative pathology confirmed the presence of residual invasive breast cancer in the breast and/or metastatic tumor lesions in axillary lymph nodes;
6. Has signed and agreed to participate in the PKUPH breast disease cohort study.

Exclusion Criteria:

1. Lack of clinical and pathological data (such as imaging data and pathological data);
2. Patients with metastatic breast cancer or bilateral breast cancer;
3. Failure to perform radical surgery;
4. Receiving other regimens besides the established neoadjuvant regimens.

The therapy choice Arm 1: The postoperative adjuvant regimen is a combination of trastuzumab and pertuzumab, with a planned treatment duration of 1 year; Arm 2: Postoperative adjuvant therapy was T-DM1, with a planned treatment duration of 1 year.

Primary end point 3-years invasive disease free survival

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients with HER2 positive breast cancer were diagnosed by biopsy in Peking University People's hospital;
* 2) The clinical stages before treatment were T1-T4, N0-N3, M0;
* 3) Received treatment and operation in our hospital, and had hospitalization records;
* 4) Receive at least 4 cycles of trastuzumab and pertuzumab target therapy combined chemotherapy as neoadjuvant therapy
* 5) Postoperative pathology confirmed the presence of residual invasive breast cancer in the breast and/or metastatic tumor lesions in axillary lymph nodes;
* 6) Has signed and agreed to participate in the PKUPH breast disease cohort study.

Exclusion Criteria:

* 1) Lack of clinical and pathological data (such as imaging data and pathological data);
* 2) Patients with metastatic breast cancer or bilateral breast cancer;
* 3) Failure to perform radical surgery;
* 4) Receiving other regimens besides the established neoadjuvant regimens.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HER2 positive breast cancer patients with residual invasive breast cancer after neoadjuvant chemotherapy combined with trastuzumab and pertuzumab
Sampling Method: Probability Sample
Enrollment: 2092 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
invasive disease free survival | 3 years
  Time from study enrollment to the first occurrence of the following events defined as failure: local recurrence of ipsilateral invasive breast cancer, contralateral invasive breast cancer, distant recurrence or death from any cause

SECONDARY OUTCOMES:
disease free survival | 3 years
  Time from study enrollment to the first occurrence of the following events defined as failure, including ipsilateral local recurrence, contralateral breast cancer, distant recurrence or death from any cause
distant disease free survival | 3 years
  Time from study enrollment to distant recurrence and metastasis
breast cancer specific survival | 3 years
  Time from study enrollment to death due to breast cancer
overall survival | 3 years
  Time from study enrollment to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: shu wang, doctor, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China